CLINICAL TRIAL: NCT07119931
Title: A Single-Arm, Single-Center, Phase II Clinical Study Evaluating the Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Iparomlimab and Tuvonralimab Injection Plus Bevacizumab in Patients With Initially Potentially Resectable Hepatocellular Carcinoma (ITBHaic Study)
Brief Title: A Clinical Study Evaluating HAIC Combined With Iparomlimab and Tuvonralimab Injection Plus Bevacizumab in Patients With Initially Potentially Resectable Hepatocellular Carcinoma (ITBHaic Study)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2025-0126
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HCC
Keywords: lparomlimab and Tuvonralimab Injection; HAIC; bevacizumab
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lparomlimab and Tuvonralimab Injection in Combination with HAIC and bevacizumab (Experimental): lparomlimab and Tuvonralimab Injection in Combination with HAIC and bevacizumab
  Interventions: Drug: lparomlimab and Tuvonralimab Injection in Combination with HAIC and bevacizumab

INTERVENTIONS:
Drug: lparomlimab and Tuvonralimab Injection in Combination with HAIC and bevacizumab — Iparomlimab and Tuvonralimab Injection（Q1706）: 7.5 mg/kg, q3w, given on Day 1 (±7 days) of each 21-day cycle; Bevacizumab: 7.5 mg/kg, q3w, administered on Day 1 (±7 days) of each 21-day cycle; HAIC:Oxaliplatin 85 mg/m² via arterial infusion over 2-3 hours, Levoleucovorin 200 mg/m² via arterial infusion over 1-2 hours, 5-Fluorouracil 400 mg/m² via arterial bolus injection, followed by continuous arterial infusion of 2400 mg/m² over 23 hours, q3w, with the treatment interval not exceeding 4 weeks.

SUMMARY:
Major Objectives To evaluate the efficacy of HAIC combined with Iparomlimab and Tuvonralimab injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) plus bevacizumab as a conversion therapy in patients with potentially resectable HCC, assessed by the conversion resection rate.

DETAILED DESCRIPTION:
This single-center, single-arm, phase II clinical study aims to evaluate the efficacy and safety of HAIC combined with Iparomlimab and Tuvonralimab injection (QL1706, an Anti-PD-1/CTLA-4 Combined Antibody) plus bevacizumab in patients with potentially resectable HCC. The study consists of four periods: screening, treatment, safety follow-up, and survival follow-up.Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily join this study, sign the informed consent form, and demonstrate good compliance;
2. Age ≥ 18 years, regardless of gender;
3. HCC confirmed histologically/cytologically or meeting the clinical diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2024 Edition), with no evidence of extrahepatic metastasis;
4. Potentially resectable HCC must meet ALL of the following criteria:

   a. Deemed unsuitable for primary surgical resection at the current stage by the Multidisciplinary Team (MDT) assessment at the research center; b. At least one untreated measurable lesion according to RECIST v1.1 criteria. (Note: Subjects who received prior local therapy for non-target lesions are eligible. Local therapy must have been completed at least 4 weeks prior to baseline scans.); c. Largest tumor diameter ≥5 cm AND ≤3 tumor lesions; d. Absence of Vp3-Vp4 stage portal vein tumor thrombus (PVTT) as per the Japanese PVTT classification system; e. Oligometastasis is permitted;
5. No prior systemic therapy for HCC (including investigational systemic agents);
6. Child-Pugh score class A or well-compensated class B (score ≤7);
7. Subjects with HBV or HCV infection must meet the following criteria:

1) HBV-infected subjects (HBsAg positive or HBV-DNA positive): Must have received guideline-recommended antiviral therapy for at least 3 days prior to the first study treatment, demonstrating a decreasing trend in HBV-DNA levels. Must continue to receive standard antiviral therapy throughout the study period; 2) HCV-infected subjects (HCVAb positive or HCV RNA positive): Must be in a stable condition per investigator assessment. If receiving antiviral therapy, must continue treatment throughout the study period; 3) Co-infection with HBV and HCV is not allowed. (Note: A history of HCV infection with undetectable HCV-RNA is considered absence of current HCV infection); 8.ECOG Performance Status score of 0-1 (Appendix 1); 9.Life expectancy ≥3 months; 10.Adequate organ function within 7 days prior to treatment, meeting all the following criteria: Hemoglobin (Hb) ≥90 g/L; White blood cell count (WBC) ≥3.5 × 10⁹/L; Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; Platelet count (PLT) ≥75 × 10⁹/L; AST and ALT ≤5 × upper limit of normal (ULN); Total bilirubin ≤3 × ULN; Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance (CrCl) ≥40 mL/min (Appendix 2); Urinalysis showing urine protein <2+(For subjects with baseline urinalysis showing urine protein ≥2+, a 24-hour urine collection must demonstrate 24-hour urine protein <1 g); Adequate coagulation function, defined as: International Normalized Ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5 × ULN; Normal thyroid function, defined as: Thyroid-stimulating hormone (TSH) within normal range. (Subjects with baseline TSH outside normal range may enroll if free triiodothyronine (FT3) or total T3 and free thyroxine (FT4) are within normal limits); 11.Male subjects and subjects of childbearing potential must use highly effective contraception from informed consent signing until 6 months after last study treatment. Subjects of childbearing potential must have a negative pregnancy test within 7 days prior to first treatment.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Histologically/cytologically confirmed HCC containing fibrolamellar, sarcomatoid, or cholangiocarcinoma components;
3. History of other primary malignancies within 5 years (except adequately treated and stable non-melanoma skin cancer, basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix);
4. Current or prior central nervous system (CNS) metastases or leptomeningeal metastasis;
5. Bleeding tendency, high bleeding risk, or coagulation dysfunction: including but not limited to thromboembolic events (e.g., cerebrovascular accident, deep vein thrombosis, pulmonary embolism) within 6 months prior to screening; and/or history of hemoptysis (≥2.5 ml bright red blood per episode) within 3 months prior to screening; current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for treatment; significant risk of gastrointestinal bleeding as judged by the investigator;
6. Presence of unhealed fractures, wound dehiscence requiring intervention, wound healing complications; tracheoesophageal fistula, gastrointestinal perforation or fistula, or intra-abdominal abscess within 6 months prior to screening;
7. Major surgery within 4 weeks before first dose (defined as Grade III or higher surgical procedures, excluding central venous catheter placement, tumor biopsy, etc.) or significant trauma with incomplete recovery;
8. Significant cardiovascular diseases (e.g., NYHA Class II or higher heart failure, myocardial infarction, or cerebrovascular events within 3 months before initiating study treatment), unstable arrhythmias, or unstable angina;
9. Active autoimmune diseases or history of autoimmune disorders including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, hypophysitis, vasculitis, systemic lupus erythematosus; Note: Excludes hypothyroidism stabilized with physiologic hormone replacement, type I diabetes controlled with stable insulin therapy, or autoimmune thyroiditis managed with stable hormone replacement.
10. Diagnosed immunodeficiency or anticipated need for systemic immunosuppressive therapy during study treatment, or prior use of systemic corticosteroids/immunosuppressants before first treatment; Note: Excludes topical/nasal/inhaled corticosteroids, physiologic systemic corticosteroids (≤10 mg/day prednisone equivalents), and transient corticosteroid use for COPD/asthma/allergy prophylaxis;
11. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia on screening chest CT scan;
12. Severe infection within 4 weeks before initiating study treatment, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks before first dose (excluding antiviral therapy for HBV/HCV);
13. Poorly controlled comorbidities despite optimal management before first treatment: Uncontrolled hyperglycemia (defined as fasting blood glucose ≥7 mmol/L, unstable oral hypoglycemic regimen, or unstable glycemic control per specialist assessment); Uncontrolled hypertension (SBP >150 mmHg and/or DBP >100 mmHg after ≥2 antihypertensive agents) or history of hypertensive crisis/encephalopathy; Refractory malignant pleural effusion, ascites, or pericardial effusion (defined as symptomatic re-accumulation requiring re-intervention within 2 weeks after drainage);
14. Known hypersensitivity to the investigational drug or its excipients;
15. Any other severe/uncontrolled comorbidity that may compromise safety or efficacy assessments per investigator judgment (e.g., hepatic encephalopathy, uncorrectable coagulopathy, hepatorenal syndrome, or cachexia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Conversion resection rate | up to 12 month
  The percentage of initially unresectable patients who underwent curative resection after protocol-specified conversion therapy.

SECONDARY OUTCOMES:
R0 Resection Rate | up to 12 month
  Proportion of patients achieving complete tumor resection with microscopically negative margins after successful conversion therapy
Pathological Complete Response | up to 12 month
  The proportion of patients in whom no residual viable tumor cells are detected upon histopathological examination of the surgically resected specimen.
Major Pathological Response | up to 12 month
  the proportion of patients with significantly reduced residual viable tumor cells in the surgically resected specimens (typically defined as ≤50% residual viable tumor cells, according to the Chinese Expert Consensus on Conversion and Perioperative Therapy for Primary Liver Cancer (2024 Edition)).
Objective response rate | up to 12 month
  the percentage of participants in the analysis population who had a CR(Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) usingRECIST1.1 based oninvestiqator assessment
Disease Control Rate | up to 12 month
  DCR was defined as the percentage of participants in the analysis population whohave CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) orSD (Neither sufficient shrinkage for PR nor sufficient increase for PD lat ≥20% increase in targetlesion SOD and absolute SOD increase of >5 mm.
Duration of Response | up to 12 month
  For participants who demonstrated a confirmed CR (disappearance of all targetlesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigatorassessment, DOR was defined as time from first documented CR or PR until PD or deathwhichever occurs first.
Progression-Free Survival (PFS) | up to 12 month
  PFS was defined as the time from first dose of study treatment to the firstdocumented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whicheveroccurred first.
Recurrence-Free Survival | up to 36 month
  The time from treatment initiation to the first recurrence or death from any cause, whichever occurs first.
Time To Progression | up to 12 month
  the time from randomization to disease progression per investigator-assessed RECIST 1.1. Death without progression will be censored at last tumor assessment.
Overall survival | up to 36 month
  OS was defined as the time from the first dose of study drug to death due to anycause.
Time To Deterioration | up to 12 month
  the time from treatment initiation to first deterioration (i.e., a ≥10-point decrease from baseline in the EORTC QLQ-C30 global score).
Symptom Improvement Rate | up to 12 month
  the number of subjects with "improvement" (≥10-point decrease in symptom score from baseline) achieving best overall response divided by the number of subjects with baseline symptom score ≥10;

IPD SHARING:
Plan to Share IPD: No